CLINICAL TRIAL: NCT05054361
Title: Crosstalk Between Mucosal-Associated Invariant T Cells and the Gut Microbiota and Mucosa in the Development of Type 1 Diabetes in Children
Brief Title: Crosstalk Between Mucosal-Associated Invariant T (MAIT) Cells and the Gut Microbiota and Mucosa in the Development of Type 1 Diabetes in Children
Acronym: MAIT-DT1
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); Tampere University (Other); Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: C19-47; 2020-A00312-37 (Other: N° ID RCB)
Record Dates: First submitted 2021-06-08; First posted 2021-09-23 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Type1diabetes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, stools, urines and gut mucosa samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- recent onset patients: patients with recently diagnosed type 1 diabetes
  Interventions: Diagnostic Test: MAIT cells analysis; Diagnostic Test: MAIT cytokines production analysis; Diagnostic Test: Lactulose/Mannitol Test; Procedure: UGI Endoscopy; Diagnostic Test: Coxsackie virus B infection status
- at risk patients: patients with a high genetic risk type 1 diabetes
  Interventions: Diagnostic Test: MAIT cells analysis; Diagnostic Test: MAIT cytokines production analysis; Diagnostic Test: Lactulose/Mannitol Test; Diagnostic Test: Coxsackie virus B infection status
- control subjects: control patients (no risk of type 1 diabetes and no diagnosed type 1 diabetes)
  Interventions: Diagnostic Test: MAIT cells analysis; Diagnostic Test: MAIT cytokines production analysis; Diagnostic Test: Lactulose/Mannitol Test; Diagnostic Test: Coxsackie virus B infection status
- control subjects for endoscopy: patients without type 1 diabetes requiring UGI endoscopy for any medical reason
  Interventions: Diagnostic Test: MAIT cells analysis; Diagnostic Test: MAIT cytokines production analysis; Procedure: UGI Endoscopy; Diagnostic Test: Coxsackie virus B infection status

INTERVENTIONS:
Diagnostic Test: MAIT cells analysis — For FACS analysis, MAIT cells will be identified as CD3+ CD4- CD161high Vα7.2+ T cells. Surface markers will be analyzed to determine their activation status (CD25, CD69, CD44), their exhaustion (PD1, KLRG1, TIM3), their migration capacity (CCR6), and their proliferation and survival will be analyzed by Ki67 and BCL2 expression.
Diagnostic Test: MAIT cytokines production analysis — Cytokine production will be assessed after PMA-ionomycin activation, followed by intracytoplasmic staining with antibodies against IL-2, IFN-γ TNF-α, IL-2, IL-4, IL-10, IL-13, IL-17 and granzyme B. To determine the capacity of MAIT cells to response to TCR stimulation (exhaustion), in vitro stimulation will be performed in the presence of specific bacterial ligands. Activation marker expression will be analyzed by FACS and cytokines released in the supernatant by Cytometry based assay.
Diagnostic Test: Lactulose/Mannitol Test — After an overnight fast, the patients will drink 50 ml solution of 5 g lactulose and 2 g mannitol. Urine will be collected during before and 5 hours later.
  Groups: at risk patients; control subjects; recent onset patients
Procedure: UGI Endoscopy — Duodenal biopsy collection and analysis. Biopsies will be analyzed by qPCR for the expression of key epithelial molecules such as the fucosyl transferase 2 (fut2), tight junction proteins (occludin, claudin4), antimicrobial peptides (Reg3, LL37) and mucus component (mucin 2). Immune cells function will also be assessed by q-PCR for key cytokines/molecules such as IL-23, IL-17, IL-22, Foxp3, IL-10, TGFb and CVB.
  Groups: control subjects for endoscopy; recent onset patients
Diagnostic Test: Coxsackie virus B infection status — Serology against CVB and CVB specific-qPCR measurement in gut microbiota samples will be performed in all patients of the three cohorts, and analysis of the gut mucosa by qPCR and immunochemistry with anti-CVB VP1 protein mAb will be performed on a subset of patients.
Diagnostic Test: Coxsackie virus B infection status — Stool samples are collected and directly kept under anaerobic condition. Within an hour the samples are processed: one fraction is aliquoted and frozen at -80°C and another fraction is used to prepared fecal supernatant for the bioassay of MAIT ligands, aliquoted and frozen. Bioassay to measure the presence of MAIT cell ligands by bioassays using WT3 cell line as well as plate bound MR117. 16S sequencing of all samples and according to the results obtained with the bioassay and 16S, 10 samples will be selected for metagenomic analysis.

SUMMARY:
To investigate in a prospective way changes in Mucosal-Associated Invariant T (MAIT) cells frequency, phenotype and function in link with the gut microbiota, gut integrity and the presence of Coxsackie virus B in two cohorts of pediatric patients: patients with a high genetic risk of type 1 diabetes and pediatric patients with recently diagnosed T1D by comparison with control subjects

Tasks:

1. To measure blood MAIT cells frequency, phenotype and function in the three cohorts
2. To analyze gut microbiota and the presence of Coxsackie B enterovirus (CVB) and their impact on MAIT cell function
3. To evaluate gut integrity and analyze the gut mucosa
4. To integrate all the data obtained with T1D development and evolution

DETAILED DESCRIPTION:
Subjects: Multi study. Subjects will be included in the pediatric diabetes and endocrinology unit in Necker Sick children hospital and in the pediatric unit of ANTONY hospital.

* Recent-onset (RO) n=40: New onset patients will be included shortly after diagnosis.
* At risk (AR) cohort n=70: Routinely screened siblings of T1D patients previously tested positive for HLA DR3 and DR4 will be asked to be a part of the study.
* Control (C) cohort (n=50): Control subjects will be patients consulting at Necker Hospital for endocrine testing
* Control for Endoscopy (CE) n= 20: patients consulting at Necker Hospital or at Antony hospital for UGI endoscopy

Analysis:

MAIT cell analysis: For FACS analysis, MAIT cells will be identified as CD3+ CD4- CD161high Vα7.2+ T cells. Surface markers will be analyzed to determine their activation status (CD25, CD69, CD44), their exhaustion (PD1, KLRG1, TIM3), their migration capacity (CCR6), and their proliferation and survival will be analyzed by Ki67 and BCL2 expression. Cytokine production will be assessed after PMA-ionomycin activation, followed by intracytoplasmic staining with antibodies against IL-2, IFN-γ TNF-α, IL-2, IL-4, IL-10, IL-13, IL-17 and granzyme B. To determine the capacity of MAIT cells to response to TCR stimulation (exhaustion), in vitro stimulation will be performed in the presence of specific bacterial ligands. Activation marker expression will be analyzed by FACS and cytokines released in the supernatant by Cytometry based assay.

Gut microbiota analysis: Stool samples are collected and directly kept under anaerobic condition. Within an hour the samples are processed: one fraction is aliquoted and frozen at -80°C and another fraction is used to prepared fecal supernatant for the bioassay of MAIT ligands, aliquoted and frozen. Bioassay to measure the presence of MAIT cell ligands by bioassays using WT3 cell line as well as plate bound MR117. 16S sequencing of all samples and according to the results obtained with the bioassay and 16S, 10 samples will be selected for metagenomic analysis.

Coxsackie virus B (CVB) infection status: Specific antibodies against coxsackie virus B and CVB specific-qPCR measurement in gut microbiota samples will be performed in all patients of the three cohorts, and analysis of the gut mucosa by q-PCR and immunochemistry will be performed on a subset of patients.

Gut integrity: the investigators will assess the permeability of the intestine using the Lactulose-Mannitol test in a sub sample of RO, RD and AR groups (> 5 years of age, n=20). In brief after an overnight fast, the patients will drink 50 ml solution of 5 g lactulose and 2 g mannitol. Urine will be collected during before and 5 hours after ingestion.

Gut mucosa analysis: In a subset of patients (without celiac disease as determined by the dosage of antibodies against transglutaminase), duodenal biopsies will be obtained during an IUG endoscopy . Duodenal biopsy will be performed in RD subjects older than 8 years of age and in CE subjects older than 4 years of age. These biopsies will be analyzed by qPCR for the expression of key epithelial molecules such as the fucosyl transferase 2 (fut2), tight junction proteins (occludin, claudin4), antimicrobial peptides (Reg3, LL37) and mucus component (mucin 2). Immune cells function will also be assessed by q-PCR for key cytokines/molecules such as IL-23, IL-17, IL-22, Foxp3, IL-10, TGFb and CVB.

Based on previous study, the sample size should allow statistical differences between AR, RO and C groups. The investigators anticipate to observe blood MAIT cell abnormalities in RO patients and some at risk children after seroconversion but before diabetes onset. This new data will strengthen our predictive model (see preliminary data). Since MAIT cells recognize bacterial ligand we hypothesize that MAIT cells alteration could occur in parallel with microbiota changes and/or CVB infection. The investigators anticipate observing gut mucosa abnormalities in RO children and the severity of these abnormalities may correlate with the level of MAIT cells defect and the presence of CVB infection. The investigators expect to demonstrate that MAIT cells represent a new biomarker of progression toward diabetes as well as a functional immune marker of the aggressiveness of the autoimmune disease. As such this study could determine the accurate therapeutic window for preventive strategies based on MAIT cells manipulation.

ELIGIBILITY:
Inclusion Criteria:

Recent onset group

* age > 12 months and < 15 years
* recently diagnosed type 1 diabetes according ISPAD criteria

At risk subjects:

* age > 12 months and < 15 years
* siblings of type 1 diabetic patient
* HLA DR3 and DR4 positive

Control subjects:

* age > 12 months and < 15 years
* no HLA associated with high risk type 1 diabetes
* no antibodies against pancreas antigenes

Control subjects for UGI endoscopy:

* age > 12 months and < 15 years
* suspicion of coeliac disease or gastritis

Exclusion Criteria:

For all groups:

* no health care insurance
* parents or tutors unable to sign the consent
* personal history of autoimmune disease and/or inflammatory disease except from T1D for RD and CE groups
* use of corticosteroids during the month before inclusion
* pregnant subjects
* medical contraindication of anesthetic topics

For control subjects for UGI endoscopy control and Recent onset-endoscopy group:

* age below 8 years for Recent onset-endoscopy group
* age below 4 for UGI endoscopy control group
* cardiac or respiratory insufficiency, cardiac rhythm disorders, coagulation disease, patients treated with anticoagulant or antiaggregant drug
* history of allergy to anesthetic drug

Ages: 12 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Study population: patients recently diagnosed with type 1 diabetes and patients with a high risk of type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-08-11 (Estimated); Study Completion 2027-08-14 (Estimated)

PRIMARY OUTCOMES:
blood MAIT cells frequency | Sample collected the day of enrollment (Control group and at risk patients) or up to 7 days after diagnosis and day of enrollment (recent onset group)
  percentage of MAIT cells in the peripheral blood

SECONDARY OUTCOMES:
MAIT cells membrane markers analysis | Sample collected the day of enrollment (Control group and at risk patients) or up to 7 days after diagnosis and day of enrollment (recent onset group)
  CD25 positive cells in percentage, CD69 positive cells in percentage, CD44 positive cells in percentage, PD1 positive cells in percentage , KLRG1 positive cells in percentage, TIM3 positive cells in percentage
Cytokines production in the cytoplasm of the MAIT | Sample collected the day of enrollment (Control group and at risk patients) or up to 7 days after diagnosis and day of enrollment (recent onset group)
  Antibodies against IL- 2 , IFN-y, TNF-α, IL-2, IL-10, IL-13, IL-17 and granzyme B expressed in Cells %
MAIT cell ligands measurements | Sample collected the day of enrollment (Control group and at risk patients) or up to 7 days after diagnosis and day of enrollment (recent onset group)
  Percentage of MAIT cells activated in vitro when cultivated in presence of subject stool sample
Presence of CVB in the stools | Sample collected the day of enrollment (Control group and at risk patients) or up to 7 days after diagnosis and day of enrollment (recent onset group)
  CVB specific ARN detection in subjects stools samples by qPCR
Blood immunoglobulins against CVB infection statu | Sample collected the day of enrollment (Control group and at risk patients) or up to 7 days after diagnosis and day of enrollment (recent onset group)
  Specific antibodies (Ig G) against CVB measurements in patients blood sample
Measurement of intestinal gut mucosal permeability | Sample collected the day of enrollment (Control group and at risk patients) or up to 7 days after diagnosis and day of enrollment (recent onset group)
  Assessing the permeability of the intestine using the Lactulose-Mannitol test. Concentration of lactulose and manitol in subjects urine samples in mg/dl
Evaluation of gut mucosal integrity | Sample collected the day of enrollment (Control group and at risk patients) or up to 7 days after diagnosis and day of enrollment (recent onset group)
  qPCR for the expression of key epithelial molecules and cytokines on gut samples
16 S sequencing in the Subjects stools | Sample collected the day of enrollment (Control group and at risk patients) or up to 7 days after diagnosis and day of enrollment (recent onset group)
  The 16S rRNA gene sequencing will be used for the classification and identification of microbes species in subjects stools. Each species will be identified and quantified as a percentage of the total number of identified species in the stools.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hopital privé d'Antony, Antony
  - Hopital Necker enfants malades, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rouxel O, Da Silva J, Beaudoin L, Nel I, Tard C, Cagninacci L, Kiaf B, Oshima M, Diedisheim M, Salou M, Corbett A, Rossjohn J, McCluskey J, Scharfmann R, Battaglia M, Polak M, Lantz O, Beltrand J, Lehuen A. Cytotoxic and regulatory roles of mucosal-associated invariant T cells in type 1 diabetes. Nat Immunol. 2017 Dec;18(12):1321-1331. doi: 10.1038/ni.3854. Epub 2017 Oct 9. PMID 28991267
- [Background] Rouland M, Beaudoin L, Rouxel O, Bertrand L, Cagninacci L, Saffarian A, Pedron T, Gueddouri D, Guilmeau S, Burnol AF, Rachdi L, Tazi A, Mouries J, Rescigno M, Vergnolle N, Sansonetti P, Christine Rogner U, Lehuen A. Gut mucosa alterations and loss of segmented filamentous bacteria in type 1 diabetes are associated with inflammation rather than hyperglycaemia. Gut. 2022 Feb;71(2):296-308. doi: 10.1136/gutjnl-2020-323664. Epub 2021 Feb 16. PMID 33593807